CLINICAL TRIAL: NCT06141902
Title: The Effects of Jing Si Herbal Tea on Physical and Psychological Symptoms in Peripheral Blood Hematopoietic Stem Cell Donors
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB111-125-A; IMAR-111-01-17 (Other Grant/Funding Number: BuddhistTCGH)
Record Dates: First submitted 2023-11-05; First posted 2023-11-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-10

CONDITIONS: Pain Syndrome; Emotional Stress
MeSH Terms: conditions — Somatoform Disorders; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NORMAL (Other): daily diet
  Interventions: Other: Jing Si Herbal Drink
- Take Jing Si Herbal Drink (No Intervention): Take Jing Si Herbal Drink daily

INTERVENTIONS:
Other: Jing Si Herbal Drink — Jing Si Herbal Drink
  Arms: NORMAL

SUMMARY:
This study aim to explore the impact of Jing Si Herbal Tea on pain and emotional stress in peripheral blood stem cell donors.

ELIGIBILITY:
Inclusion Criteria:

* health Men or women aged 20 to 55 years old
* willing to take Jing Si Herbal Drink

Exclusion Criteria:

* no willing to take Jing Si Herbal Drink;
* Previously already take Jing Si Herbal Drink daily

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in pain assessed by questionnaires | 5 day
  For each of the pain sites includes: headache、bone、joint & muscle, indicate the severity of present using the following scale (baseline vs. follow-up).
  grade 0: fully active, able to carry on all pre-disease performance without restriction
  grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work
  grade 2: ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours
  grade 3: capable of only limited self-care, confined to bed or chair more than 50% of waking hours
  grade 4: completely disabled, cannot carry on any self-care, totally confined to bed or chair
  grade 5: dead

SECONDARY OUTCOMES:
Changes in anxiety assessed by questionnaires | 21 days
  Difference in donor Health State Trait Anxiety Index (STAI) scores (baseline vs. follow-up).
  The STAI questionnaire consists of 20 items for assessing "state anxiety" and 20 items for assessing "trait anxiety," with a raw score of 20 to 60 points for each scale.
  The state anxiety scale evaluates the current state of anxiety associated with a special situation, measuring subjective feelings of apprehension, tension, nervousness, worry, and activation of the autonomic nervous system, whereas the trait anxiety scale evaluates proneness to anxiety .
  The level of anxiety was determined according to the percentile rank obtained using the raw score of each questionnaire and was classified as low anxiety (1st-23th percentile), moderate anxiety (25th75th percentile) and high anxiety (77th-99th percentile).

CONTACTS AND LOCATIONS:
Locations (1):
- Hualiien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City, Taiwan